CLINICAL TRIAL: NCT05395637
Title: Reliability of Longshi Scale With Remote Assessment of Smartphone Video Calls for Stroke Patients'Activities of Daily Living
Brief Title: Reliability of Longshi Scale With Remote Assessment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220224002
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Telemedicine
Keywords: Stroke; Tele-rehabilitation; Activities of Daily Living
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assessed with the remote assessment of Longshi Scale first and then with bedside assessment
- Assessed with the bedside assessment of Longshi Scale first and then with remote assessment

SUMMARY:
To explore the reliability of remote Longshi Scale assessment with smartphone video calls by comparing the consistency of remote assessment and bedside assessment, as well as the test-retest reliability of the remote assessment. The evaluation duration of these two methods was recorded and the level of satisfaction of patients and evaluators was investigated.

ELIGIBILITY:
Inclusion Criteria:

* a.Stroke survivors

  1. aged 18 and above;
  2. diagnosed with cerebral infraction or intracerebral hemorrhage;
  3. stroke onset2 weeks;
  4. stable vital signs (heart rate, blood pressure, respiratory rate, oxygen saturation and temperature);
  5. voluntary or guardian consent to participate in the study.

     b.Evaluators

  <!-- -->

  1. registered rehabilitation practitioner;
  2. experience in rehabilitation scientific research or education related work for more than two years

Exclusion Criteria:

* a.Stroke survivors

  1. brain tumor, Parkinson's disease or active epilepsy within past three months;
  2. a history of mental illness such as mania or delirium;
  3. participation in any other clinical study. b.Evaluators

  <!-- -->

  1. unable to finish the training of Longshi Scale or use smartphones proficiently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors from the Department of Rehabilitation Medicine at Shenzhen Second People's Hospital are invited to participate in this study according to the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Consistency of the disability degree evaluated using the remote assessment and the bedside assessment of Longshi Scale. | Within 24 hours
  Weighted kappa(wK) and Bland-Altman were used to determined the consistency between the results of remote assessment method and bedside assessment method. The interpretation of wK scores was in accordance with published standards (values>0.75 indicating excellent agreement beyond chance; 0.4~0.75, moderate agreement beyond chance; <0.4, poor agreement beyond chance).

SECONDARY OUTCOMES:
The test-retest reliability of the remote video assessment | Within 24 hours after first evaluation
  the result of remote assessment test-retest was analyzed by Weighted kappa(wK) scores.The interpretation of wK scores was in accordance with published standards (values>0.75 indicating excellent agreement beyond chance; 0.4~0.75, moderate agreement beyond chance; <0.4, poor agreement beyond chance).
Satisfaction survey of remote assessment | Within 24 hours after the remote assessment
  The satisfaction survey data were summarized as mean±standard deviation, and also summarized as the percentage of satisfaction categories.
Assessment duration | Within 24 hours
  The assessment duration was analyzed by independent t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China